CLINICAL TRIAL: NCT02917837
Title: Effect of a Diagnostic Imaging Utilization Report on Family Physician Ordering Practices in the Eastern Health Regional Health Authority, Newfoundland and Labrador
Brief Title: Effect of Diagnostic Imaging Utilization Reports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: NL SUPPORT Strategy for Patient-Oriented Research (Unknown)
Responsible Party: Principal Investigator, Kris Aubrey-Bassler, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NLSUPPORT-Aubrey
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Diagnostic Imaging Utilization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual QCNL report group (Active Comparator): Physicians receive the usual Quality of Care Newfoundland and Labrador utilization report: This reports ranks the physician on a figure of their peers according to the total number of tests ordered in a one-year period.
  Interventions: Other: Usual QCNL DI utilization report
- Usual QCNL report plus detailing. (Experimental): This group receives the usual QCNL report described above. Shortly after the reports are sent, this group will be contacted at least three times to attempt to arrange a single in-person detailing session.
  Interventions: Other: Usual QCNL DI utilization report; Other: Detailing
- New utilization report (Experimental): This group will receive a new type of report that shows individual physician ordering per 100 patients compared to the mean of all physicians, adjusted for patient complexity (age, sex, comorbidity, education, income, rurality).
  Interventions: Other: New DI utilization report
- New utilization report plus detailing (Experimental): New type of report plus detailing as described above.
  Interventions: Other: New DI utilization report; Other: Detailing

INTERVENTIONS:
Other: Usual QCNL DI utilization report — See arm descriptions.
  Arms: Usual QCNL report group; Usual QCNL report plus detailing.
Other: New DI utilization report — See arm descriptions.
  Arms: New utilization report; New utilization report plus detailing
Other: Detailing — In-person detailing, usually with a small group of family physicians and a peer (physician) facilitator to discuss the topic over a 30-60 minute period.
  Arms: New utilization report plus detailing; Usual QCNL report plus detailing.

SUMMARY:
Diagnostic imaging (DI) tests (for example, x-ray tests, ultrasounds, CT scans, or MRIs) are used by health care providers to help diagnose patient illness, but decisions regarding when these tests should be ordered are subjective. As a result, some physicians order these tests more than others. Ordering rates between clinicians seeing similar kinds of patients have been shown to be considerably different, suggesting that many of the tests are unnecessary. DI currently accounts for about 6.6% of Canadian hospital budgets, but this percentage may be much higher in Newfoundland where test ordering rates are almost twice the national average. However, cost is not the only concern. Over-testing can lead to further unnecessary testing to follow-up on harmless findings, and in the case of CT, large doses of potentially harmful radiation. We suspect that many clinicians are not aware that they order more DI tests than their peers. We will therefore develop a "report card" for family physicians in the province that shows them how many tests they are ordering compared to other physicians in the region. We expect that physicians who are over-ordering DI tests will reduce the number of tests they order after receiving their report cards. This is a low-cost way to potentially prevent expensive over-ordering of DI tests that can easily be implemented in the province's other health regions and elsewhere. The Quality of Care Newfoundland and Labrador (QCNL) organization in the province currently provides feedback reports and in-person detailing sessions to physicians, but the effectiveness of these interventions has not been studied.

DETAILED DESCRIPTION:
The purpose of this trial is to compare the effectiveness of two versions of a DI utilization feedback report for family physicians, and determine whether in-person detailing sessions offer additional benefit in changing ordering practices. Group practices (i.e. all physicians practicing at the same address) of family physicians and general practitioners will be stratified by community of practice within Eastern Health, then randomized into one of four groups: 1. A usual QCNL feedback report alone, 2. A usual QCNL feedback report plus in-person detailing, 3. A new feedback report alone, 4. A new feedback report plus in-person detailing. Communities with fewer than five physicians will be grouped with similar communities for stratified randomization purposes.

Physicians will be provided a semi-annual (every 6 months) report card outlining the number of CT scans, ultrasounds and plain x-rays they ordered per 100 patients for whom they were the primary provider. We will assume that the primary provider is the most frequent biller of primary care services. Participants will receive a link to the report card via email from the Newfoundland and Labrador Medical Association (NLMA) by a two-step process: The initial email gives a brief description of the report and contains a link which then redirects the clinician to a secure web page that displays the individual clinician diagnostic imaging utilization in a prior one year period compared to the aggregate of their peers in the same region. Physicians in the detailing groups will be contacted to arrange a single in-person session with one of their colleagues to discuss the detailing reports.

ELIGIBILITY:
There are no restrictions on the age of participants.

Inclusion Criteria:

* 1) All family physicians or general practitioners practicing within Eastern Health. In order to obtain an accurate assessment of the report in real-world implementation, we are requesting the right to enroll everyone who meets the inclusion criteria, and to waive the requirement to obtain informed consent
* 2) Be the most frequent provider of primary care billings for a minimum of 20 patients during the period.

Exclusion Criteria:

* 1) Physicians who will be within the Eastern Health network for a relatively short period, e.g. clinicians engaged in an exchange program for training, or locums.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Combined CT, x-ray and ultrasound exam orders per patient | 1 year
  Number of DI tests ordered per patient seen

SECONDARY OUTCOMES:
Clinician subgroup Diagnostic imaging exam orders per patient | 1 year
  Clinicians will be divided into high and low test ordering subgroups (based on pre-intervention ordering practices). The primary outcome will be measured in these subgroups as a secondary outcome.
Uptake of detailing | 1 year
  Proportion of invited physicians who take part in a detailing session
CT exam orders per patient | 1 year
X-ray exam orders per patient | 1 year
Ultrasound exam orders per patient | 1 year
Uptake of utilization reports | 1 year
  Proportion of physicians in report groups who open the link for the online report.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Aubrey-Bassler, MD, CCFP(EM), Principal Investigator — Primary Healthcare Research Unit, Memorial University
Locations (1):
- Health Sciences Centre, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Background] Mittal MK, Zorc JJ, Garcia-Espana JF, Shaw KN. An assessment of clinical performance measures for pediatric emergency physicians. Am J Med Qual. 2013 Jan-Feb;28(1):33-9. doi: 10.1177/1062860612443849. Epub 2012 Jun 7. PMID 22679126
- [Background] Jain S, Elon LK, Johnson BA, Frank G, Deguzman M. Physician practice variation in the pediatric emergency department and its impact on resource use and quality of care. Pediatr Emerg Care. 2010 Dec;26(12):902-8. doi: 10.1097/PEC.0b013e3181fe9108. PMID 21088636
- [Background] Goldzweig CL, Orshansky G, Paige NM, Miake-Lye IM, Beroes JM, Ewing BA, Shekelle PG. Electronic health record-based interventions for improving appropriate diagnostic imaging: a systematic review and meta-analysis. Ann Intern Med. 2015 Apr 21;162(8):557-65. doi: 10.7326/M14-2600. PMID 25894025
- [Background] Jain S, Frank G, McCormick K, Wu B, Johnson BA. Impact of Physician Scorecards on Emergency Department Resource Use, Quality, and Efficiency. Pediatrics. 2015 Sep;136(3):e670-9. doi: 10.1542/peds.2014-2363. Epub 2015 Aug 10. PMID 26260722
- [Background] Schwappach DL, Blaudszun A, Conen D, Ebner H, Eichler K, Hochreutener MA. 'Emerge': Benchmarking of clinical performance and patients' experiences with emergency care in Switzerland. Int J Qual Health Care. 2003 Dec;15(6):473-85. doi: 10.1093/intqhc/mzg078. PMID 14660530
- [Background] Campbell SM, Reeves D, Kontopantelis E, Sibbald B, Roland M. Effects of pay for performance on the quality of primary care in England. N Engl J Med. 2009 Jul 23;361(4):368-78. doi: 10.1056/NEJMsa0807651. PMID 19625717
- [Background] Campbell S, Reeves D, Kontopantelis E, Middleton E, Sibbald B, Roland M. Quality of primary care in England with the introduction of pay for performance. N Engl J Med. 2007 Jul 12;357(2):181-90. doi: 10.1056/NEJMsr065990. No abstract available. PMID 17625132
- [Background] Michie S, Johnston M, Abraham C, Lawton R, Parker D, Walker A; "Psychological Theory" Group. Making psychological theory useful for implementing evidence based practice: a consensus approach. Qual Saf Health Care. 2005 Feb;14(1):26-33. doi: 10.1136/qshc.2004.011155. PMID 15692000
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Klabunde CN, Harlan LC, Warren JL. Data sources for measuring comorbidity: a comparison of hospital records and medicare claims for cancer patients. Med Care. 2006 Oct;44(10):921-8. doi: 10.1097/01.mlr.0000223480.52713.b9. PMID 17001263